CLINICAL TRIAL: NCT02070679
Title: Efficacy of Vitamin E in Preventing Contrast-Induced Acute Kidney Injury Following Coronary Angiography
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Urmia University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Chancellor of research, Mir Hossein Seyyed-Mohammadzad, Urmia University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UMSU-Cardiology-1
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Stable Angina; Unstable Angina; Non ST Segment Elevation Myocardial Infarction; Post MI
Keywords: Alpha-tocopherol; Vitamin E; Contrast-Induced Acute Kidney Injury; Coronary angiography
MeSH Terms: conditions — Angina, Stable; Angina, Unstable | interventions — Vitamin E; alpha-Tocopherol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
- Vit-E (Active Comparator): 600 IU on 12 hours before angiography and 400 IU on 2 hours before angiography
  Interventions: Drug: Vitamin E

INTERVENTIONS:
Drug: Vitamin E
  Other Names: Alpha-tocopherol
  Arms: Vit-E

SUMMARY:
The purpose of this study is to evaluate the effect of vitamin E on preventing from incidence of contrast induced acute kidney injury (CI-AKI) in the patients who undergone coronary angiography.

ELIGIBILITY:
Inclusion Criteria:

1. All patients whon have either stable coronary artery disease (CAD) or recent acute coronary disease (ACS) and are scheduled for coronary angiography.
2. Patients who have eGFR ≤60 ml/min/1.73 m2

Exclusion Criteria:

1. Allergy to contrast media
2. Cardiogenic shock
3. Pulmonary edema
4. Overt cardiac failure or left ventricular ejection fraction ≤ 30%
5. Acute kidney injury
6. The history of receiving contrast media for any medical diagnostic or therapeutic procedures during previous 5 days
7. The history of dialysis
8. Being pregnant
9. Having recent acute myocardial infarction
10. Taking antioxidants and nephrotoxic drugs including NSAID and ACE-I on previous 2 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2014-02; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The development of CI-AKI in group receiving vitamin E compared with placebo | Within 72 hours after coronary angiography

SECONDARY OUTCOMES:
Changes in the serum level of Cr and the amount of eGFR | Within 72 hours

CONTACTS AND LOCATIONS:
Locations (2):
- Iran (2):
  - Seyyed-al-Shohada Heart Center, UMSU, Urmia, West Azerbaijan Province
  - Taleghani Hospital, UMSU, Urmia, West Azerbaijan Province

REFERENCES:
- [Derived] Rezaei Y, Khademvatani K, Rahimi B, Khoshfetrat M, Arjmand N, Seyyed-Mohammadzad MH. Short-Term High-Dose Vitamin E to Prevent Contrast Medium-Induced Acute Kidney Injury in Patients With Chronic Kidney Disease Undergoing Elective Coronary Angiography: A Randomized Placebo-Controlled Trial. J Am Heart Assoc. 2016 Mar 15;5(3):e002919. doi: 10.1161/JAHA.115.002919. PMID 27068631